CLINICAL TRIAL: NCT07267390
Title: MOVIE-TRACE Study: Investigating MPXV Viral Clearance in Mpox Cases and Secondary Attack Rate in Contacts
Brief Title: Investigating MPXV Viral Clearance in Mpox Cases and Secondary Attack Rate in Contacts
Acronym: MOVIE-TRACE
Status: Recruiting | Type: Observational
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: University of Kinshasa (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Oriol Mitja, Associate Professor, Infectious Diseases and Global Health, Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Other Study IDs: MOVIE-TRACE
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Mpox (Monkeypox)
Keywords: viral clearance; secondary attack rate; DRC
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, lesion swap, oropharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MOVIE: Mpox confirmed case
- TRACE: Contact of a MOVIE case

SUMMARY:
The MOVIE-TRACE project includes two complementary observational studies designed to improve the understanding of Mpox virus infection and its transmission within affected communities. The MOVIE study aims to describe the dynamics of viral clearance in patients with confirmed Mpox. It measures how the viral load changes over time in different biological samples to inform decisions about patient management and isolation guidelines. The TRACE study focuses on understanding how mpox spreads from confirmed cases to their contacts. It will estimate the Secondary Attack Rate (SAR) and identify factors associated with transmission risk. The results will help guide public health strategies for contact tracing, vaccination, and outbreak control.

DETAILED DESCRIPTION:
Starting in late 2023, an increasing number of confirmed cases of Mpox caused by clade I Mpox virus (MPXV) were reported across several provinces of the Democratic Republic of the Congo (DRC). In August 2024, the World Health Organization (WHO) declared the ongoing outbreak a Public Health Emergency of International Concern due to its expanding geographic spread and significant public health impact.

Mpox is transmitted through direct contact with skin or mucosal lesions of infected individuals, contaminated materials. MPXV can be detected in multiple biological samples, including skin lesion swabs, blood, throat swabs, and occasionally urine. However, there is still limited information on how long and in which compartments the virus can persist, as well as on how efficiently it spreads between individuals during community outbreaks caused by clade I virus.

The MOVIE-TRACE project includes two complementary observational studies designed to address these critical gaps in knowledge and to strengthen the understanding of clade I MPXV infection in the DRC.

The MOVIE study aims to describe how MPXV is cleared from the body over time among patients with PCR-confirmed Mpox infection. Despite the importance of isolation and infection control in outbreak management, there is limited evidence on how long individuals remain infectious. MOVIE addresses this critical gap by conducting longitudinal follow-up of Mpox-positive patients for up to two months, with several scheduled visits during which multiple biological specimens are collected. These samples will be analyzed to assess viral persistence in different body compartments and to characterize the kinetics of viral clearance. The findings will help refine isolation duration, improve clinical management, and guide infection prevention policies.

The TRACE study seeks to understand how Mpox spreads from confirmed cases to their contacts. By systematically collecting exposure data and testing contacts for infection, TRACE will estimate the Secondary Attack Rate (SAR) and identify factors that increase the likelihood of transmission. This information will support public health measures such as contact tracing, quarantine strategies, and targeted vaccination in endemic regions.

Together, MOVIE and TRACE will generate essential evidence on both viral clearance and transmission of clade I MPXV, providing a comprehensive understanding of the infection and informing data-driven outbreak response strategies in the Democratic Republic of the Congo.

ELIGIBILITY:
Inclusion Criteria:

* MOVIE Study:

  * Individuals of any sex and age presenting with lesions clinically suggestive of Mpox, as assessed by a trained health worker.
  * Symptom onset within the 10 days prior to the baseline assessment.
  * Willingness and ability to comply with study procedures and attend scheduled follow-up visits for up to two months.
  * Availability for follow-up throughout the study period.
  * Provision of written informed consent by the participant, or consent by a legally authorized representative for minors or individuals unable to provide it themselves.
  * Assent obtained from children aged 12 years or older.
  * For participants who cannot read or write, witnessed consent will be obtained.
* TRACE Study:

  * Individuals who have had close physical contact with a polymerase chain reaction (PCR)-confirmed Mpox case within 14 days from the onset of symptoms in the index case.
  * Close physical contact is defined as being within 2 meters of an infected person-particularly in enclosed spaces-for at least 5 minutes (based on CDC's 2-meter rule for droplet transmission).
  * Willingness and ability to comply with the study protocol and attend scheduled follow-up assessments.
  * Provision of written informed consent by the participant, or consent by a legally authorized representative for individuals unable to provide it themselves.

Exclusion Criteria:

* MOVIE Study:

  * Cases of severe Mpox requiring hospitalization.
  * Individuals with a confirmed alternative diagnosis explaining their illness.
  * Prior vaccination against Mpox.
  * Individuals over 40 years of age who report having received smallpox vaccination during infancy.
* TRACE Study:

  * Prior vaccination against Mpox.
  * Individuals over 40 years of age who report having received smallpox vaccination during infancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with confirmed Mpox infection, regardless of age or sex.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Viral clearance in skin lesions | From day 1 to day 56
  Time to undetectable MPXV viral load (>35 Ct) in skin lesions (Number of days)
Viral clearance in oropharyngeal swabs | From day 1 to day 56
  Time to undetectable MPXV viral load (>35 Ct) in oropharyngeal swabs (Number of days)
Viral clearance in blood | From day 1 to day 56
  Time to undetectable MPXV viral load (>35 Ct) in blood (Number of days)
Mpox transmission among cases and their contacts | From day 1 to day 14
  Estimation of Secondary Attack Rate (SAR)

SECONDARY OUTCOMES:
Factors of transmission | From day 1 to day 14
  Identification of factors linked to transmission

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Mitjà, Professor, Principal Investigator — Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia
Locations (1):
- Univeristy of Kinshasa, Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be shared under reasonable request

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT07267390/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT07267390/ICF_001.pdf